CLINICAL TRIAL: NCT03379051
Title: Phase I/II Study of Venetoclax or Lenalidomide in Combination With Ublituximab and Umbralisib in Subjects With Relapsed or Refractory CLL/SLL and NHL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic/Business Decision
Sponsor: TG Therapeutics, Inc. (Industry)
Collaborators: James P. Wilmot Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U2-VEN-109
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Chronic Lymphocytic Leukemia; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — venetoclax; umbralisib; ublituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ublituximab + Umbralisib + Venetoclax (Experimental): Ublituximab at a fixed IV infusion dose Days 1, 8 and 15 followed by maintenance infusions TGR-1202 oral daily dose Venetoclax oral daily dose
  Interventions: Drug: Venetoclax; Drug: Umbralisib; Biological: Ublituximab
- Ublituximab + Umbralisib + Lenalidomide (Experimental): Ublituximab at a fixed IV infusion dose Days 1, 8 and 15 followed by maintenance infusions; Umbralisib and Lenalidomide both administered days 1 - 21 of every 28 days
  Interventions: Drug: Umbralisib; Biological: Ublituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Venetoclax — BCL-2 Inhibitor
  Other Names: Venclexta
  Arms: Ublituximab + Umbralisib + Venetoclax
Drug: Umbralisib — PI3K-Delta Inhibitor
  Other Names: TGR-1202
Biological: Ublituximab — Glycoengineered Anti-CD20 mAb
  Other Names: TG-1101
Drug: Lenalidomide — Thalidomide Analog, immunomodulatory agent with antiangiogenic and antineoplastic properties
  Other Names: Revlimid
  Arms: Ublituximab + Umbralisib + Lenalidomide

SUMMARY:
Phase I/II Study of Venetoclax or Lenalidomide in Combination with Ublituximab and Umbralisib in Subjects with Relapsed or Refractory CLL/SLL and NHL

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of B-cell Chronic Lymphocytic Leukemia, or Non-Hodgkin's Lymphoma
* Refractory to or relapsed after at least 1 prior treatment regimen
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Known hepatitis B virus, hepatitis C virus or HIV infection
* Known histological transformation from CLL to an aggressive lymphoma (Richter's)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Determine Acceptable Adverse Events That Are Related to Treatment | 12 months

SECONDARY OUTCOMES:
Overall Response and Complete Remission Rate | 12 months
Minimum Residual Disease (MRD) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Barr, MD, Study Chair — Wilmot Cancer Institute - University of Rochester
Locations (3):
- United States (3):
  - TG Therapeutics Investigational Trial Site, Chicago, Illinois
  - TG Therapeutics Investigational Trial Site, Rochester, New York
  - TG Therapeutics Investigational Trial Site, Cleveland, Ohio

REFERENCES:
- [Derived] Hill BT, Ma S, Zent CS, Baran AM, Wallace DS, Advani A, Winter A, Winter J, Gordan L, Karmali R, Liesveld JL, Mulford DA, Rowland C, Bui A, Sportelli P, Miskin HP, Weiss MS, Friedberg JW, Barr PM. Response-adapted, time-limited venetoclax, umbralisib, and ublituximab for relapsed/refractory chronic lymphocytic leukemia. Blood Adv. 2024 Jan 23;8(2):378-387. doi: 10.1182/bloodadvances.2023010693. PMID 37871300